CLINICAL TRIAL: NCT02322346
Title: Peritonsillar Infiltration With Levobupivacaine for Relief of Posttonsillectomy Pain: Does Concentration Have Any Effect?
Brief Title: Peritonsillar Infiltration With Levobupivacaine for Posttonsillectomy Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Sanem Cakar Turhan, Specialist, Ankara University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 134-3866
Record Dates: First submitted 2014-12-13; First posted 2014-12-23 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Pain
Keywords: posttonsillectomy pain; levobupivacaine
MeSH Terms: conditions — Pain | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group S (Placebo Comparator): Preincisional bilateral peritonsillar infiltration of a total of 6 mL of saline
  Interventions: Other: Group S
- Group LL (Active Comparator): Preincisional bilateral peritonsillar infiltration of levobupivacaine 0.25% (3 mL to each tonsil).
  Interventions: Drug: Group LL
- Group HL (Active Comparator): Preincisional bilateral peritonsillar infiltration of levobupivacaine 0.5% (3 mL to each tonsil).
  Interventions: Drug: Group HL

INTERVENTIONS:
Other: Group S — Peritonsillar infiltration with saline Additional remifentanil 1 µgr kg-1 IV was administered to the patients if HR was increased by 25 % of the basal value.
  During postoperative period, symptoms such as pain, fever and dysphagia, adverse affects such as nausea and vomiting and hemorrhage were evaluated. Pain was evaluated by FLACC (Faces, leg, activity, cry, consolability), FPRS (Faces pain rating scale) ve Wong-Baker facies scales at postoperative 0, 30 and 60 minutes and 2, 6, 12 and 24 hours. Total analgesic consumption during the postoperative period were recorded. If the patients had no complication, they were discharged at the postoperative 24th hour.
  Other Names: Saline
  Arms: Group S
Drug: Group LL — Peritonsillar infiltration with low-dose of levobupivacaine 0.25%. Additional remifentanil 1 µgr kg-1 IV was administered to the patients if HR was increased by 25 % of the basal value.
  During postoperative period, symptoms such as pain, fever and dysphagia, adverse affects such as nausea and vomiting and hemorrhage were evaluated. Pain was evaluated by FLACC (Faces, leg, activity, cry, consolability), FPRS (Faces pain rating scale) ve Wong-Baker facies scales at postoperative 0, 30 and 60 minutes and 2, 6, 12 and 24 hours. Total analgesic consumption during the postoperative period were recorded. If the patients had no complication, they were discharged at the postoperative 24th hour.
  Other Names: Chirocaine 0.25%
  Arms: Group LL
Drug: Group HL — Peritonsillar infiltration with high dose of levobupivacaine 0.5%. Additional remifentanil 1 µgr kg-1 IV was administered to the patients if HR was increased by 25 % of the basal value.
  During postoperative period, symptoms such as pain, fever and dysphagia, adverse affects such as nausea and vomiting and hemorrhage were evaluated. Pain was evaluated by FLACC (Faces, leg, activity, cry, consolability), FPRS (Faces pain rating scale) ve Wong-Baker facies scales at postoperative 0, 30 and 60 minutes and 2, 6, 12 and 24 hours. Total analgesic consumption during the postoperative period were recorded. If the patients had no complication, they were discharged at the postoperative 24th hour.
  Other Names: Chirocaine 0.5%
  Arms: Group HL

SUMMARY:
The investigators aimed to evaluate the effects of different concentrations of preincisional peritonsillar levobupivacaine (0.25% ve 0.5%) on postoperative pain and bleeding

DETAILED DESCRIPTION:
72 ASA I-II patients between 3 and 12 years of age who scheduled to undergo tonsillectomy were enrolled in this randomized, prospective and placebo-controlled study. The indications for tonsillectomy were recurrent infections and tonsillar hypertrophy leading to obstructive symptoms.

The patients included to the study were randomly assigned to one of the 3 groups to receive different concentrations of levobupivacaine or saline.

The mean arterial pressure (MAP) and heart rates (HR) of all patients were recorded during the whole anesthesia and surgical procedures. The duration of anesthesia and surgery were also recorded. Additional remifentanil 1 µgr kg-1 IV was administered to the patients if HR was increased by 25 % of the basal value.

During postoperative period, symptoms such as pain, fever and dysphagia, adverse affects such as nausea and vomiting and hemorrhage were evaluated. Pain was evaluated by FLACC (Faces, leg, activity, cry, consolability), FPRS (Faces pain rating scale) ve Wong-Baker facies scales at postoperative 0, 30 and 60 minutes and 2, 6, 12 and 24 hours. Total analgesic consumption during the postoperative period were recorded. If the patients had no complication, they were discharged at the postoperative 24th hour.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 3 and 12 who were scheduled to undergo tonsillectomy due to recurrent infections leading to obstructive symptoms
* Patients aged 3 and 12 who were scheduled to undergo tonsillectomy due to tonsillar hypertrophy leading to obstructive symptoms.

Exclusion Criteria:

* Hypersensitivity to sevoflurane, benzodiazepine, fentanyl analogues, propofol and components, paracetamol, levobupivacaine
* Presence of coagulation disorders and chronic diseases
* Presence of regular use of analgesics
* Presence of analgesic use within 24 hours prior to surgery
* Presence of upper respiratory system infection
* Inability to understand the pain scales, being unable to communicate.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Change in postoperative pain | 24 hours
  pain assessed with FPRS (Faces pain rating scale)

SECONDARY OUTCOMES:
Presence of dysphagia | 24 hours
  number of participants with dysphagia and without dysphagia.

CONTACTS AND LOCATIONS:
Overall Officials: K.Sanem Cakar Turhan, Specialist, Principal Investigator — Ankara University

REFERENCES:
- [Derived] Cakar Turhan KS, Salviz EA, Beton S, Timuroglu ST, Catav S, Ozatamer O. Peritonsillar infiltration with levobupivacaine for posttonsillectomy pain relief: does concentration have any effect? A double-blind randomized controlled clinical study. Eur Rev Med Pharmacol Sci. 2015 Apr;19(7):1276-84. PMID 25912590